CLINICAL TRIAL: NCT02615730
Title: A Phase Ib/IIa, Open-Label, Dose Finding Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of PI3Kβ Selective Inhibitor (GSK2636771) Administered in Combination With Paclitaxel in Advanced Gastric Adenocarcinoma
Brief Title: PI3Kβ Selective Inhibitor With Paclitaxel, Advanced Gastric Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0204
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — GSK2636771; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel & GSK2636771 (Experimental): Increasing dose levels of GSK2636771 (300 mg or 400 mg once daily) in combination with a fixed dose of paclitaxel (80 mg/m2 on Days 1, 8 and 15 of a 28-day treatment cycle)
  Interventions: Drug: GSK2636771; Drug: Paclitaxel

INTERVENTIONS:
Drug: GSK2636771 — Increasing dose levels of GSK2636771 (300 mg or 400 mg once daily)
Drug: Paclitaxel — fixed dose of paclitaxel (80 mg/m2 on Days 1, 8 and 15 of a 28-day treatment cycle)

SUMMARY:
This is a Phase Ib/IIa, open-label, non-randomized, dose-escalation, multi-center study to evaluate the safety, tolerability, pharmacokinetics (PK), and clinical activity of oral GSK2636771 in combination with intravenous (IV) paclitaxel in two independent subject populations: subjects with PTEN-deficient, advanced gastric adenocarcinoma.

DETAILED DESCRIPTION:
This is a Phase Ib/IIa, open-label, non-randomized, dose-escalation, multi-center study to evaluate the safety, tolerability, pharmacokinetics (PK), and clinical activity of oral GSK2636771 in combination with intravenous (IV) paclitaxel in two independent subject populations: subjects with PTEN-deficient, advanced gastric adenocarcinoma. This study will be conducted in two phases: the Dose Escalation Phase and the Dose Expansion Phase. The Dose Escalation Phase (Phase Ib) is designed to determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D) of GSK2636771 administered in combination with paclitaxel. The Dose Expansion Phase (Phase IIa) will further evaluate the safety and clinical activity of the RP2D as determined in the Dose Escalation Phase.

ELIGIBILITY:
Inclusion criteria:

1. histologically or cytologically confirmed diagnosis of advanced gastric adenocarcinoma
2. Has a PTEN-deficient tumor as documented from archival or fresh (from biopsy) tumor tissue or has shown genomic alterations in PI3K pathway genes (PIK3CB, PI3KR1, PTEN, etc.) as assessed in a local laboratory.
3. Has had no prior taxane exposure (preferred) or at least 6 months since last taxane exposure.
4. Eastern Cooperative Oncology Group performance status of 0 or 1
5. measurable or evaluable disease as determined by RECIST 1.1.
6. Is able to swallow and retain orally administered medication
7. adequate baseline organ function

Exclusion criteria

1. prior treatment with any AKT, mammalian target of rapamycin (mTOR) inhibitors or PI3K pathway inhibitors
2. Has any unresolved Grade 2 (per CTCAE v4.0) toxicity from previous anti-cancer therapy at the time of enrollment such as neuropathy, except alopecia or Grade 2 anemia (if hemoglobin is ≥9.0 g/dL)
3. Has CNS metastases
4. Has a QTc interval >450 msec or QTc >480 msec for subjects with bundle branch block (BBB)
5. Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2636771 or hypersensitivity to drug formulated in polyoxyl 35 castor oil, NF such as paclitaxel.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II dose | 4 weeks
  Recommended Phase II dose for phase 1
Progression-free survival | 6 weeks
  Progression-free survival for phase 2

SECONDARY OUTCOMES:
Dose limiting toxicity | 28 days
  Dose limiting toxicity for phase 1

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, Principal Investigator — Yonsei Cancer Center
Locations (1):
- Severance Hospital, Yonsei University Health System, Yonsei Cancer Center, Seoul, South Korea